CLINICAL TRIAL: NCT07004387
Title: Perioperative Use of Amino Acids in Recipients of Orthotopic Liver Transplantation as a Renal Protective Factor
Acronym: PAATHO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Dr Sotero del Rio (Other)
Responsible Party: Principal Investigator, GUILLERMO MOLINA MANCERO, SPECIALIST IN INTENSIVE CARE MEDICINE, Hospital Dr Sotero del Rio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AMUCI-25
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Hepatic Failure; Liver Transplant; Renal Failure, Acute
Keywords: liver transplant; renal failiure; amino acids; surguery; ICU
MeSH Terms: conditions — Liver Failure; Acute Kidney Injury | interventions — amino-acid, glucose, and electrolyte solution; Arginine

STUDY DESIGN:
Intervention Model Description: A pilot, prospective, non-randomized, analytical study with intervention, in which adult patients scheduled for orthotopic liver transplantation will be assigned to receive an intravenous infusion of a mixture of amino acids including L-arginine, at a dose of 2 g per kg of ideal body weight up to a maximum of 100 g per day, from their admission to the operating room until three days after the surgery. The infusion will begin in the operating room, prior to the start of the surgery, and will be performed through an exclusive lumen of a central venous catheter (CVC) immediately after the CVC is in place; the infusion will continue when the patient is in the intensive care unit (ICU); as soon as the patient begins enteral nutrition, the infusion will be reduced to meet the 2 g per kg of protein intake per day, up to a maximum of 100 g per day, until completing 72 hours of infusion. The control group consists of cases of previously transplanted patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amino acid interventión group (Experimental): Patients over 18 years old scheduled to undergo liver transplantation who are expected to have an ICU stay of at least 24 hours in the immediate postoperative period, regardless of the cause of liver failure and whether it was stable liver failure or acute on chronic liver failure. They will receive an intravenous infusion of a mixture of amino acids that includes L-arginine, at a dose of 2 g per kg of ideal body weight up to a maximum of 100 g per day, from their admission to the operating room until three days after the surgery.
  Interventions: Drug: Amino acid solution; Drug: Amino Acid infusion

INTERVENTIONS:
Drug: Amino acid solution — Adult patients scheduled for orthotopic liver transplant to receive an intravenous infusion of a mixture of amino acids including L arginine, at a dose of 2 g per kg of ideal body weight up to a maximum of 100 g per day, from their admission to the operating room until three days after surgery; the infusion will begin in the operating room prior to the start of the surgery, will be administered through an exclusive lumen of a central venous catheter (CVC) immediately after the CVC is in place; the infusion will continue when the patient is in the intensive care unit (ICU); as soon as the patient begins enteral nutrition, the infusion will be reduced to meet the dose of 2 g per kg of protein intake per day up to a maximum of 100 g daily, until completing 72 H of infusion. The Control Group consists of previously transplanted patients at this institution who did not receive this type of therapy.
  Other Names: l arginine
Drug: Amino Acid infusion — adult patients scheduled for orthotopic liver transplant to receive an intravenous infusion of a mixture of amino acids including L arginine, at a dose of 2 g per kg of ideal body weight up to a maximum of 100 g per day, from their admission to the operating room until three days after surgery; the infusion will begin in the operating room prior to the start of the surgery, will be administered through an exclusive lumen of a central venous catheter (CVC) immediately after the CVC is in place; the infusion will continue when the patient is in the intensive care unit (ICU); as soon as the patient begins enteral nutrition, the infusion will be reduced to meet the dose of 2 g per kg of protein intake per day up to a maximum of 100 g daily, until completing 72 H of infusion. The Control Group consists of previously transplanted patients at this institution who did not receive this type of therapy.
  Other Names: l arginina

SUMMARY:
Orthotopic liver transplantation is the definitive treatment for end-stage liver failure, with renal failure being an important complication of this procedure that has implications for long- and short-term prognosis, affecting ICU stay and hospitalization time. Several studies have suggested that intravenous amino acids, particularly L-arginine, may have protective effects on renal function due to increased renal blood flow, which could be explained by enhanced production of nitric oxide among other mechanisms that are still unclear. In this context, we developed the hypothesis that the infusion of an amino acid solution in the perioperative period could reduce the incidence of acute renal failure in this group of patients; for this, we conducted a monocentric, analytical, prospective, interventional pilot study comparing standard treatment (in historically transplanted patients) with a group of patients who were administered amino acids in the perioperative period, considering that this medication is low-cost and has practically minimal side effects.

DETAILED DESCRIPTION:
The primary objectives will be to measure the occurrence of acute kidney injury according to KDIGO criteria, evaluate the behavior of BUN and creatinine, as well as the initiation and duration of renal replacement therapy if necessary, use of vasopressors, diuresis, liver enzymes and bilirubin, lactate; this will be during the first 10 days postoperatively. Additionally, as a secondary objective, to measure all-cause mortality at 30 days. The study protocol must be approved by the institution's ethics committee. The treatment with amino acids will be carried out using Aminoven 10% from Fresenius Kabi available at the hospital. Fresenius Kabi has not had and will not have any role in the conception, development, data collection, and/or tabulation of data and/or publication of the results of this study. Data collection will be undertaken by specific personnel chosen from among those healthcare providers of liver transplantation, surgery, anesthesiology, and intensive care services.

ELIGIBILITY:
Inclusion Criteria:

* All patients assigned to receive a liver transplant will be evaluated for eligibility.
* Patients over 18 years old scheduled for a liver transplant will be considered eligible if it is expected that they will have an ICU stay of at least 24 hours in the immediate postoperative period, regardless of the cause of liver failure and whether it was stable liver failure or acute on chronic liver failure.
* They must have a baseline measurement of serum creatinine that does not exceed 30 days prior to surgery or can be taken before the transplant surgery.

Exclusion Criteria:

* Patients under 18 years old will be excluded.
* Patients with a need for chronic hemodialysis, patients with chronic kidney disease with an estimated glomerular filtration rate of less than 30 ml per minute per 1.73 square meters of body surface area calculated by the Cockcroft-Gault equation.
* Patients with acute renal failure requiring acute intermittent or continuous renal replacement therapy during the hospitalization for surgery.
* Patients who refuse informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-27 (Estimated); Primary Completion 2026-05-27 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
acute kidney failiure | During the first 10 days of the postoperative period
  measure the incidence of renal failure in the postoperative period of liver transplantation

SECONDARY OUTCOMES:
liver function post Liver Transplant | For ten days after the postoperative period
  serial measurement of liver enzymes and bilirubin, lactate.
Need for vasopressors | For ten days postoperatively.
  Doses of noradrenaline, adrenaline, and/or vasopressin
Mortality from all causes. | At 28 days
  Mortality from all causes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sotero Del Rio, Santiago, Puente ALTO, Chile

IPD SHARING:
Plan to Share IPD: Undecided
REQUIRES NEW REVIEW BY THE ETHICS COMMITTEE

REFERENCES:
- [Background] Landoni G, Monaco F, Ti LK, Baiardo Redaelli M, Bradic N, Comis M, Kotani Y, Brambillasca C, Garofalo E, Scandroglio AM, Viscido C, Paternoster G, Franco A, Porta S, Ferrod F, Calabro MG, Pisano A, Vendramin I, Barucco G, Federici F, Severi L, Belletti A, Cortegiani A, Bruni A, Galbiati C, Covino A, Baryshnikova E, Giardina G, Venditto M, Kroeller D, Nakhnoukh C, Mantovani L, Silvetti S, Licheri M, Guarracino F, Lobreglio R, Di Prima AL, Fresilli S, Labanca R, Mucchetti M, Lembo R, Losiggio R, Bove T, Ranucci M, Fominskiy E, Longhini F, Zangrillo A, Bellomo R; PROTECTION Study Group. A Randomized Trial of Intravenous Amino Acids for Kidney Protection. N Engl J Med. 2024 Aug 22;391(8):687-698. doi: 10.1056/NEJMoa2403769. Epub 2024 Jun 12. PMID 38865168
- [Background] Pu H, Doig GS, Heighes PT, Allingstrup MJ, Wang A, Brereton J, Pollock C, Chesher D, Bellomo R. Intravenous amino acid therapy for kidney protection in cardiac surgery patients: A pilot randomized controlled trial. J Thorac Cardiovasc Surg. 2019 Jun;157(6):2356-2366. doi: 10.1016/j.jtcvs.2018.11.097. Epub 2018 Dec 15. PMID 30685166
- [Background] Pruna A, Losiggio R, Landoni G, Kotani Y, Redaelli MB, Veneziano M, Lee TC, Zangrillo A, Gaudino MFL, Bellomo R; for Protection Study group. Amino Acid Infusion for Perioperative Functional Renal Protection: A Meta-analysis. J Cardiothorac Vasc Anesth. 2024 Dec;38(12):3076-3085. doi: 10.1053/j.jvca.2024.08.033. Epub 2024 Aug 22. PMID 39384419
- [Background] Hoffmann K, Buchler MW, Schemmer P. Supplementation of amino acids to prevent reperfusion injury after liver surgery and transplantation--where do we stand today? Clin Nutr. 2011 Apr;30(2):143-7. doi: 10.1016/j.clnu.2010.09.006. Epub 2010 Oct 20. PMID 20965621